CLINICAL TRIAL: NCT02827838
Title: Pilot Study to Evaluate the Anti-Tumor Effect of Durvalumab (Medi4736) in Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN), Human Papilloma Virus (HPV) Positive Versus Negative, When Treated Before Surgery
Brief Title: Durvalumab Before Surgery in Treating Patients With Oral Cavity or Oropharynx Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study closed prior to meeting enrollment goal and funding issues
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00038877; NCI-2016-00639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 60116 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-07-11 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Human Papillomavirus Infection; Stage I Oral Cavity Squamous Cell Carcinoma; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Oral Cavity Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Oral Cavity Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Oral Cavity Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, surgery) (Experimental): Patients receive durvalumab IV over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot clinical trial studies how well durvalumab before surgery works in treating patients with oral cavity or oropharynx cancer. Monoclonal antibodies, such as durvalumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the effect of durvalumab on local and systemic immune activation by HPV status in patients with oral cavity and oropharynx head and neck squamous cell carcinoma (HNSCC).

II. To examine the effects of durvalumab on systemic immune response to HPV and tumor associated antigens.

III. To examine the effects of durvalumab on immune regulatory mechanisms. IV. To explore the association between levels of immune-regulatory micro-ribonucleic acid (miR) in plasma and saliva and immune response.

SECONDARY OBJECTIVES:

I. Investigate the effect of the treatment with durvalumab on the computed tomography (CT) scan and positron emission tomography (PET) scan response.

II. Evaluate the safety of a short induction treatment with durvalumab.

OUTLINE:

Patients receive durvalumab intravenously (IV) over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.

After completion of study treatment, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HNSCC of the oral cavity (OC; more than 90% patients have HPV negative cancer) or oropharynx (about 60-80% of patient have HPV positive cancer)
* Presence of radiologically of clinically documented disease. All radiology studies must be performed within 28 days prior to registration
* Any stage, considered candidates for surgery and planned for surgery either by robotic or by standard surgical technique
* Documentation of HPV tested by polymerase chain reaction (PCR) (resulted or pending)
* Willing to provide consent for an additional tissue biopsy for research purposes, to allow a part of their surgical tumor tissue to be utilized for research (in case tumor tissue has not already been saved in the tumor tissue bank), and to donate samples of blood and saliva collected weekly through the treatment
* All patients must have provided informed consent for correlative studies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Patients must have no prior exposure to immune-mediated therapy, including anti- cytotoxic T-lymphocyte protein 4 (CTLA-4), anti-programmed cell death 1, anti-programmed cell death 1 ligand 1 (PD-L1), or anti-programmed cell death ligand 2 antibodies, excluding therapeutic anticancer vaccines
* At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as > or = 10 mm in the longest diameter (except lymph nodes, which must have a short axis > or = 15 mm) with CT or magnetic resonance imaging (MRI) or clinical measurement and that is suitable for accurate repeated measurements as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines
* Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of registration, and that wound healing has occurred
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 9.0 g/dL
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) (institutional upper limit of normal)
* Total bilirubin is less than or equal to ULN, except the case in which the elevated total bilirubin is not a sign of liver disease, such as the Gilbert Syndrome, in which case a Total Bilirubin less than or equal to 2X ULN is acceptable.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: >= 60 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
* In accordance with National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) policy, protocol treatment is to begin within 2 working days of patient registration
* Written informed consent and any locally-required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States of American [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Age 18 years or older at time of study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 6 months (mo)
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* Receipt of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within the last 6 mo (before the first dose of Durvalumab).
* Mean QT interval corrected for heart rate (corrected QT [QTc]) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2) from previous anti-cancer therapy; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Active or prior documented autoimmune disease within the past 2 years; NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Patients with body weight <= 30 kg
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Durvalumab, Surgery) HPV Negative: Patients receive durvalumab IV over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.
  Durvalumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
  HPV negative
- Treatment (Durvalumab, Surgery) HPV Positive: Patients receive durvalumab IV over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.
  Durvalumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
  HPV positive
Period: Overall Study
Arm/Group | Treatment (Durvalumab, Surgery) HPV Negative | Treatment (Durvalumab, Surgery) HPV Positive
Started | 11 | 6
Completed | 11 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Durvalumab, Surgery) - HPV Negative: Patients receive durvalumab IV over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.
  Durvalumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
  HPV negative
- Treatment (Durvalumab, Surgery) - HPV Positive: Patients receive durvalumab IV over approximately 60 minutes on day 1. Treatment repeats every 2 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Within 3-17 days after last dose administration of durvalumab, patients undergo surgery. Patients may receive an additional dose of durvalumab if time to surgery is longer than 30 days.
  Durvalumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
  HPV positive
- Total: Total of all reporting groups
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.2) | 58.0 (6.5) | 58.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 5 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Immune Effector Assessed in Blood by Flow Cytometry and in Tissue by Immunohistochemistry
Description: Concentration of certain immune effector will be assessed in blood pre- and post- treatment. Descriptive statistics, confidence intervals will be calculated and 2-sample t-tests will be performed. Tumor-infiltrating immune-regulator and effector cells will be quantified (0 to 3+) using standing immunofluorescence techniques. Counts and percents will be calculated for these measures overall and by HPV (+/-) groups pre- and post-treatment. Fisher exact tests will be used to compare groups at pre- and post- treatment. Stuart-Maxwell tests (generalizations of the McNemar's Test
Time Frame: Up to 18 months
Population: This pre-specified outcome is dependent upon 1) patients having a measurable response and 2) availability of comparable cohorts of HPV positive and negative samples. Since there was a lack of measurable clinical response in all patients and the enrolled cohorts were unbalanced, the data for this outcome was not measured/evaluated and therefore is not available for analysis.
Arm/Group | Treatment (Durvalumab, Surgery)
Number analyzed (Participants) | 0

2. Primary Outcome: Immune-regulatory miR Responses as Measured in Plasma Assessed by Quantitative Reverse Transcriptase PCR (qRT-PCR)
Description: Percent change of levels of immune-regulatory miRs assessed in plasma assessed pre-treatment and one week post-treatment.
Time Frame: At baseline and at one week post treatment start
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive
Number analyzed (Participants) | 11 | 6
percent change from baseline
  miR 146 | 27.5 [-24.5 to 124.2] | 1251.6 [116.6 to 6039.3]
  miR 155 | 19.7 [-24.2 to 364.3] | 814 [100.7 to 2154.9]
  miR 181 | 25.7 [1.7 to 189.8] | 893.2 [107.8 to 3880.8]
  miR 20a | -15.6 [-55.2 to 6.4] | 520.6 [43.4 to 1226.9]
  miR 223 | 13.7 [-61.3 to 51.0] | 1031.2 [43.9 to 3034.1]
  miR 335 | 12.5 [-44.9 to 142.8] | 1166.0 [336.2 to 2070.6]
  miR 125 | 43.4 [-9.2 to 79.6] | 194.5 [4.2 to 1789.6]

3. Primary Outcome: Systemic Immune Response to HPV Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Lab results will be compared between patients who are HPV+ and HPV- using 2 sample t-tests. These measures will be compared in several ways. First, baseline, pre-treatment levels will be examined using descriptive statistics (n, mean, standard deviations, range). These measures will be examined overall and by HPV (+/-) groups. For each measure, and time point, 95% confidence intervals will be estimated. Next, two sample t-tests will be performed to compare levels of the measures at baseline. Next, measures taken post-treatment will be examined in a similar manner (descriptive statistics and 2-
Time Frame: Up to 18 months
Population: as for outcome 1
Arm/Group | Treatment (Durvalumab, Surgery)
Number analyzed (Participants) | 0

4. Primary Outcome: Regulatory Responses Assessed in Blood by Flow Cytometry and in Tissue by Immunohistochemistry
Description: Concentration of certain regulatory cells will be assessed in blood pre- and post- treatment. Descriptive statistics, confidence intervals will be calculated and 2-sample t-tests will be performed. Tumor-infiltrating immune-regulator and effector cells will be quantified (0 to 3+) using standing immunofluorescence techniques. Counts and percents will be calculated for these measures overall and by HPV (+/-) groups pre- and post-treatment. Fisher exact tests will be used to compare groups at pre- and post- treatment. Stuart-Maxwell tests (generalizations of the McNemar's Tes
Time Frame: Up to 18 months
Population: as for outcome 1
Arm/Group | Treatment (Durvalumab, Surgery)
Number analyzed (Participants) | 0

5. Primary Outcome: Immune-regulatory miR Responses as Measured in Saliva Assessed by Quantitative Reverse Transcriptase PCR (qRT-PCR)
Description: Percent change of levels of immune-regulatory miRs assessed in saliva assessed pre-treatment and one week post-treatment.
Time Frame: Baseline and one week post treatment start
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive
Number analyzed (Participants) | 11 | 6
percent change from baseline
  miR 146 | 251.3 [-12.3 to 497.9] | 105.3 [-16.2 to 362.7]
  miR 155 | 141.2 [4.6 to 970.3] | 255.0 [0.0 to 367.5]
  miR 181 | 114.4 [-35.6 to 864.6] | 232.5 [77.8 to 558.9]
  miR 20a | 163.9 [-63.1 to 1312.3] | 113.1 [58.6 to 500.0]
  miR 223 | 66.4 [-47.0 to 502.1] | 199.2 [0.0 to 465.7]
  miR 335 | 249.4 [20.2 to 628.5] | 150.2 [0.0 to 397.6]
  miR 125 | 351.6 [-34.9 to 471.6] | 64.9 [-10.8 to 457.9]

6. Primary Outcome: Immune-regulatory miR Responses as Measured in Tumor Tissue Assessed by Quantitative Reverse Transcriptase PCR (qRT-PCR)
Description: Levels of immune-regulatory miRs assessed in blood, saliva and tumor tissue will be assessed pre- and post- treatments. Descriptive statistics, confidence intervals will be calculated and 2-sample t-tests will be performed. In addition, correlations between the different methods will be examined (i.e., correlation between saliva and blood measures, saliva and tumor measures, and blood and tumor measures).
Time Frame: Up to 18 months
Population: as for outcome 1
Arm/Group | Treatment (Durvalumab, Surgery)
Number analyzed (Participants) | 0

7. Primary Outcome: Systemic Immune Response to Tumor Associated Antigens Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: as for outcome 3
Time Frame: Up to 18 months
Population: as for outcome 1
Arm/Group | Treatment (Durvalumab, Surgery)
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of Adverse Events (AEs) as Measured by CTCAE Version 4.03
Description: AEs will be coded using the Medical Dictionary for Regulatory Activities to their organ class by preferred term. Coded AEs will be displayed by frequency, severity, and relationship to treatment (durvalumab) in the safety population. In addition, summary tables will be generated for the following situations: 1) fatigue, diarrhea, nausea and skin rash; 2) Immune-mediated reactions of any grade; 3) other adverse events graded as 3 or more by CTCAE Version 4.03; 4) Durvalumab dose reductions; 5) discontinuations of treatment with durvalumab, with specification of reason for discontinuation; and 6) changes in the surgical treatment schedule. Toxicity grades Grade I (mild), Grade II (moderate), Grade III (severe), Grade IV (life threatening) and Grade V (fatal). Toxicities of greater than or equal to Grade III (except infusion reaction) are considered worse outcomes.
Time Frame: At baseline (pre-treatment), during scheduled treatment and up to the 90-day follow up period after the last dose of study drug administered, with a median of 1 month and maximum of 13 months
Measure: Number; unit: events
Groups:
- HPV -: HPV negative
- HPV +: HPV positive
Arm/Group | HPV - | HPV +
Number analyzed (Participants) | 11 | 6
events
  Acute kidney injury - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Alanine aminotransferase increased - Possible to Definitely related - Grade 2 | 1 | 0
  Alanine aminotransferase increased - Possible to Definitely related - Grade 3 | 1 | 0
  Alkaline phosphatase increased - Possible to Definitely related - Grade 1 | 2 | 0
  Alkaline phosphatase increased - Possible to Definitely related - Grade 2 | 1 | 0
  Anemia - Unrelated or Unlikely related - Grade 3 | 2 | 0
  Anorexia - Possible to Definitely relate - Grade 1 | 1 | 1
  Aspartate aminotransferase increased - Possible to Definitely related - Grade 1 | 2 | 0
  Aspartate aminotransferase increased - Possible to Definitely related - Grade 2 | 2 | 0
  Aspartate aminotransferase increased - Possible to Definitely related - Grade 4 | 1 | 0
  Blood bilirubin increased - Possible to Definitely related - Grade 1 | 2 | 0
  Blood bilirubin increased - Possible to Definitely relate - Grade 2 | 1 | 0
  Bullous dermatitis - Possible to Definitely relate - Grade 1 | 1 | 0
  Constipation - Possible to Definitely relate - Grade 1 | 1 | 1
  Constipation - Possible to Definitely relate - Grade 2 | 1 | 0
  Device related infection - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Diarrhea - Possible to Definitely relate - Grade 1 | 3 | 0
  Diarrhea - Possible to Definitely relate - Grade 3 | 1 | 0
  Diarrhea - Unrelated or Unlikely related - Grade 1 | 4 | 1
  Fatigue - Possible to Definitely relate - Grade 1 | 6 | 3
  Fatigue - Possible to Definitely relate - Grade 2 | 1 | 0
  Fatigue - Unrelated or Unlikely related - Grade 1 | 1 | 1
  Fatigue - Unrelated or Unlikely related - Grade 2 | 1 | 0
  Head soft tissue necrosis - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Hyperglycemia - Unrelated or Unlikely related - Grade 3 | 0 | 1
  Hyperglycemia - Unrelated or Unlikely related - Grade 4 | 1 | 0
  Hypermagnesemia - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Hypertension - Unrelated or Unlikely related - Grade 3 | 0 | 1
  Hypoalbuminemia - Unrelated or Unlikely related - Grade 3 | 2 | 0
  Hypocalcemia - Unrelated or Unlikely related - Grade 3 | 4 | 0
  Hypocalcemia - Unrelated or Unlikely related - Grade 4 | 1 | 0
  Hypokalemia - Unrelated or Unlikely related - Grade 3 | 3 | 0
  Hyponatremia - Unrelated or Unlikely related - Grade 3 | 4 | 0
  Hypophosphatemia - Unrelated or Unlikely related - Grade 3 | 4 | 0
  Hypotension - Unrelated or Unlikely related - Grade 3 | 2 | 0
  Hypothyroidism - Possible to Definitely relate - Grade 2 | 0 | 1
  Leukocytosis - Unrelated or Unlikely related - Grade 3 | 1 | 1
  Lipase increased - Possible to Definitely relate - Grade 3 | 0 | 1
  Malaise - Possible to Definitely relate - Grade 1 | 1 | 0
  Nausea - Possible to Definitely relate - Grade 1 | 1 | 0
  Nausea - Unrelated or Unlikely related - Grade 1 | 3 | 0
  Neck soft tissue necrosis - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Neutrophil count decreased - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Pruritus - Possible to Definitely relate - Grade 1 | 0 | 1
  Rash maculo-papular - Possible to Definitely relate - Grade 1 | 1 | 0
  Rash pustular - Possible to Definitely relate - Grade 1 | 1 | 0
  Serum amylase increased - Possible to Definitely relate - Grade 1 | 0 | 1
  Skin ulceration - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Skin ulceration - Unrelated or Unlikely related - Grade 4 | 1 | 0
  Taste alteration (dysgeusia) - Possible to Definitely relate - Grade 1 | 0 | 1
  Urine output decreased - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Urticaria - Possible to Definitely relate - Grade 1 | 0 | 1
  Weight loss - Possible to Definitely relate - Grade 1 | 1 | 1
  Wound complication - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Wound infection - Unrelated or Unlikely related - Grade 3 | 1 | 0
  Discontinuation of Durvalumab due to immune-related hepatitis | 1 | 0

9. Secondary Outcome: Standardized Uptake Value (SUV) as Measured by PET Scans
Description: Change in SUV activity as measured by PET scans from baseline to post-treatment not specific to HPV status.
Time Frame: Up to 18 months
Population: This pre-specified outcome is dependent upon 1) patients having a measurable response and 2) availability of comparable cohorts of HPV positive and negative samples. Since there was a lack of measurable clinical response in all patients and the enrolled cohorts were unbalanced, the data for this outcome was not measured/evaluated for all patients.
Measure: Mean (Standard Error); unit: change in SUV
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive
Number analyzed (Participants) | 2 | 1
change in SUV | -0.15 (1.20) | 0 (0)

10. Secondary Outcome: Tumor Diameter Assessed Using RECIST Version 1.1 Criteria
Description: Change in tumor diameters will be compared between groups (HPV +/-) pre- and post- treatment.
Time Frame: Up to 18 months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive
Number analyzed (Participants) | 11 | 6
mm | 1.0 [0.0 to 4.0] | -2.0 [-2.0 to 2.0]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events was recorded from time of signature of informed consent, throughout the treatment period and including the follow-up period (90 days after the last dose of durvalumab), with a median of 1 month and maximum of 13 months
Arm/Group | Treatment (Durvalumab, Surgery) - HPV Negative | Treatment (Durvalumab, Surgery) - HPV Positive
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/11 | 0/6
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Durvalumab, Surgery) - HPV Negative (N=11) | Treatment (Durvalumab, Surgery) - HPV Positive (N=6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Durvalumab, Surgery) - HPV Negative (N=11) | Treatment (Durvalumab, Surgery) - HPV Positive (N=6)
Anemia (Blood and lymphatic system disorders) | 6 (8) | 5 (6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0)
Edema face (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (9) | 4 (4)
Fever (General disorders) | 3 (3) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Neck edema (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other: tumor infection per treating physician (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (5) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 5 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (18) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (20) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (15) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (19) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (18) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other: skin irritation at G-tube site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other: dental extraction site inflammation (dry sockets) (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT02827838/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT02827838/ICF_000.pdf